CLINICAL TRIAL: NCT01240967
Title: An Open-Label, Multi-Center, Phase I Study To Compare the Pharmacokinetics of a Single Oral Dose of TC-5214 (S-Mecamylamine) in Subjects With Renal Impairment With Subjects With Normal Renal Function
Brief Title: To Compare the Pharmacokinetics of a Single Oral Dose of TC-5214 in Subjects With Renal Impairment and With Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None
Other Study IDs: D4130C00008
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Volunteers; Patients; Pharmacokinetics; Renal Impairment
Keywords: Phase 1; healthy volunteers; volunteers with renal impairment; pharmacokinetics; TC-5214
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: TC-5214 — Oral tablets, single dose

SUMMARY:
The purpose of this study is to compare the absorption and distribution of a single oral dose of TC-5214 in subjects with renal impairment and with subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating females 18 to 80 years old inclusive with suitable veins for cannulation or repeated venipuncture with a weight of at least 50 kg.
* Regarding renal function, subjects will be classified as either normal or as suffering from mild, moderate or severe renal impairment. Classification of renal impairment will be based using an abbreviated 4 variable Modified Diet in Renal Disease (MDRD) equations. To ensure the assessment of consistent estimated glomerular filtration rate (eGFR) using the MDRD, a single equation will be used (see Section 6.2)
* Negative screen for Human Immunodeficiency Virus and negative results for serum hepatitis B surface antigen
* Regarding renal function, subjects will be classified as either normal or as suffering from mild, moderate or severe renal impairment. Classification of renal impairment will be based using an abbreviated 4 variable MDRD equation. To ensure the assessment of consistent estimated glomerular filtration rate (eGFR) using the MDRD, a single equation will be used.

Exclusion Criteria:

* History of any clinically significant medical, neurologic or psychiatric disease or disorder (other than those previously defined as acceptable for these population) which, in the opinion of the Investigator and sponsor, may either put the subject at risk because of participation in the study, or influence the results of the subject's ability to participate in the study: This includes seizure activity and repeated episodes of major depression.
* Subjects with a history of suicide attempts in the past year and/or seen by the Investigator as having a significant history of risk of suicide or homicide, or considered at risk for suicide or homicide during the study
* Subjects with an active renal transplant (subjects who have previously received a renal transplant and are currently undergoing dialysis due to transplant failure may be enrolled)
* Any clinically significant acute illness or medical/surgical procedure within 4 weeks of the first administration of investigational product (IP) (other than those previously defined as acceptable for these population) as judged by the Investigator.
* Positive test in drugs of abuse screens (except for prescription medications, which are verified by the Investigator), or alcohol on admission to the clinic prior to the administration of the IP

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetics (PK) of a single dose of TC-5214 in subjects with renal impairment in comparison to the results in subjects with normal renal function | For Group 1, Group 2, and Group 3 blood PK samples will be collected at predose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours postdose.
The pharmacokinetics (PK) of a single dose of TC-5214 in subjects with renal impairment in comparison to the results in subjects with normal renal function | For Group 4 blood PK samples will be collected at predose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours postdose.
  If study procedures for any subjects in Group 4 are extended by 24 hours to Day 5, PK samples will be collected at predose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours postdose.

SECONDARY OUTCOMES:
The effect of hemodialysis on TC-5214 pharmacokinetics | For Group 5 blood PK samples will be collected at predose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours postdose.
Safety and tolerability variables: Adverse events and serious adverse events (including severity), vital signs, physical examinations, laboratory parameters, electrocardiograms, and the Columbia-Suicide Severity Rating Scale. | A range of 5 days -from Screening to follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Hans A Eriksson, MD, Study Director — AstraZeneca; Thomas Marbury, MD, Principal Investigator — Orlando Clinical Research Center
Locations (2):
- United States (2):
  - Research Site, Orlando, Florida
  - Research site, Minneapolis, Minnesota

REFERENCES:
- [Derived] Alverlind S, Barassin S, Dalen P, Li Y, Toler S, Eriksson H, Tummala R. Clinical pharmacokinetics of the nicotinic channel modulator dexmecamylamine (TC-5214) in subjects with various degrees of renal impairment. Clin Drug Investig. 2014 Jul;34(7):457-65. doi: 10.1007/s40261-014-0195-0. PMID 24760402
- [Derived] Xu H, Henningsson A, Alverlind S, Tummala R, Toler S, Beaver JS, Al-Huniti N. Population pharmacokinetics of TC-5214, a nicotinic channel modulator, in phase I and II clinical studies. J Clin Pharmacol. 2014 Jun;54(6):707-18. doi: 10.1002/jcph.264. Epub 2014 Jan 16. PMID 24408516
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1414&filename=CSR-D4130C00008.pdf
- See also: CSR-D4130C00008.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1414&filename=CSR-D4130C00008.pdf
- See also: D4130C00008/Clinical Study Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1414&filename=TC5214_D4130C00008_Renal_Protocol_pdf_Redacted.pdf